CLINICAL TRIAL: NCT04523935
Title: Excessive Crying in Children With Cerebral Palsy and Communication Deficits -a Fixed-sequence, Crossover Clinical Trial
Brief Title: Excessive Crying in Children With Cerebral Palsy and Communication Deficits
Acronym: ECCCPCD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sathbhavana Brain Clinic (Other)
Responsible Party: Principal Investigator, Dr.Nagabhushana Rao Potharaju, Pediatric Neurologist, Sathbhavana Brain Clinic
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ECCP
Record Dates: First submitted 2020-08-12; First posted 2020-08-24 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Cerebral Palsy; Excessive Crying; Pain
Keywords: Allodynia; Neuropathic pain; Run-in period; childhood onset dystonia; drooling; dysphagia; hyperalgesia; muscle spasticity
MeSH Terms: conditions — Cerebral Palsy; Pain; Hyperalgesia; Neuralgia; Dystonic Disorders; Sialorrhea; Deglutition Disorders; Muscle Spasticity | interventions — Fructose; Baclofen; Diazepam; Clonazepam; Trihexyphenidyl; Tetrabenazine; Gabapentin; Topiramate; Lamotrigine; Amitriptyline

STUDY DESIGN:
Intervention Model Description: There was an initial placebo run-in period. This clinical trial was a prospective, single-center, interventional, with initial placebo-control, double-blind for initial 110 days, open-label for the next 290 days, fixed-sequence, two-treatment, two-period, crossover clinical trial. The placebo run-in period (15 days) was followed by the placebo period (15 days). After a washout period (10 days), drug treatment (360 days) was started depending on the clinical findings and investigations.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The best and most reliable form of research is a double-blind, placebo-controlled study that would eliminate the power of suggestion and prevent bias when patients' outcomes are evaluated thereby improving the reliability of clinical trial results.
  Our study was double-blind initially for 110 days until the 70th day of treatment (Figure. 1, Figure. 2.). The caregiver of the participant, the research nurse, and the outcome data collecting nurse were not aware of the drug or drug combination and the dosage. There was no contact between the research nurse, the pharmacist preparing the medicines, and the outcome data collecting nurse. The caregiver of the participant was unaware of other participants' details.
  Later, it was an open-label study for 290 days because double blinding for the total period of 400 days may not serve any additional purpose but increases the dropout risk.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo-Sequence 1 (Placebo Comparator): The placebo contained fructose powder in packets identical to the medicines.
  Interventions: Other: Placebo
- Drug-Sequence 2 (Active Comparator): GABA-B agonists, muscarinic acetylcholine receptor antagonists, inhibitors of the vesicular monoamine transporter, benzodiazepines, antiepileptics, and tricyclic antidepressants were used.
  Interventions: Drug: Baclofen, Diazepam, Clonazepam, Trihexyphenidyl, Tetrabenazine, Gabapentin, Topiramate, Lamotrigine, Amitriptyline.

INTERVENTIONS:
Other: Placebo — Fructose powder identical with the drugs was used
  Other Names: Fruit sugar, levulose.
  Arms: Placebo-Sequence 1
Drug: Baclofen, Diazepam, Clonazepam, Trihexyphenidyl, Tetrabenazine, Gabapentin, Topiramate, Lamotrigine, Amitriptyline. — Drugs were used either singly or in combination guided by clinical findings and investigations.
  Other Names: Baclofen(Liofen®),Diazepam,(Valium®),Clonazepam,(Klonopin®),Trihexyphenidyl(Artane®),Tetrabenazine(Xenazine®),Gabapentin(Neurontin®),Topiramate(Topamax®),Lamotrigine(Lamictal®),Amitriptyline(Elavil®)
  Arms: Drug-Sequence 2

SUMMARY:
Management of excessive crying in children with cerebral palsy and communication deficits [ECCCPCD] was guided by the associated clinical findings and investigations.

DETAILED DESCRIPTION:
Pain treatments are frequently hit or miss, trial & error, or because of the fear of litigations, not offered at all, particularly in cerebral palsy. Pain is an under-suspected and under-diagnosed cause of ECCCPCD. It was hypothesized that pain/discomfort was responsible for ECCCPCD, and a vicious cycle of pain-spasm-pain aggravated the pain/discomfort. So, the response of ECCCPCD to treatment guided by clinical findings & investigations was studied.

There was an initial placebo run-in period. This study was a prospective, single-center, interventional, with initial placebo-control, double-blind for initial 110 days, open-label for the next 290 days, fixed-sequence, two treatment, two-period, crossover clinical trial. The placebo run-in period (15 days) was followed by the placebo period (15 days). After a washout period (10 days), drug treatment (360 days) was started depending on the clinical findings and investigations. The drugs used either singly or in various combinations were GABA-B agonists, muscarinic acetylcholine receptor antagonists, benzodiazepines, inhibitors of the vesicular monoamine transporter, antiepileptics, and tricyclic antidepressants. The outcome measure was total, and unexplained mean cry durations in hours per day. The cry duration was measured for one 10-day period while on placebo [days P6-P15], and four 10-day periods while on treatment [T61-70, T241-250, T311-320, and T351-360]. Total and unexplained mean cry durations in hours per day were calculated from 10-day measurements of cry durations. From the 251st day of therapy, the dose was reduced by 5% every week until [ECCCPCD] started to increase. This reduction of the dose was made to confirm the efficacy of drugs and to check if the dosage requirement has reduced after 250 days of treatment. This dose was maintained until the next measurement between T311 and T320. Then the dosages were adjusted as necessary. The caregivers were allowed to volunteer any additional observations of interest. Drug adverse effects were recorded.

Epidemiological data, GMFCS levels, and MAS scores were noted at the time of enrollment. Summary statistics were tabulated and plotted. Paired t-tests and Wilcoxon tests were done to study the statistical significance.

ELIGIBILITY:
1. A child with cerebral palsy under the age of 15 years and could not communicate the reason for excessive crying because of young age or global developmental delay/profound intellectual retardation.
2. Excessive crying of >7.5 hours daily for 30 consecutive days unresponsive to treatment by the pediatrician, orthopedic surgeon, gastroenterologist, and physiotherapist.
3. Minimum cry intensity for recording: If the intensity of crying was so high that the caregiver could not hear radio, TV, or another person talking to her [sitting near her], the cry duration was recorded.
4. History, clinical, and neuroimaging findings (structural MRI) were suggestive of chronic static encephalopathy.
5. Motor impairment could be explained by an insult that occurred in the developing fetal or infant brain.

Exclusion Criteria:

1. Medicines used in the study were used in the previous 30 days, and it was impossible to taper off the drugs without worsening of symptoms.
2. Excessive crying due to known causes.
3. Progressive encephalopathies.

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 131 (Actual)
Dates: Start 2005-12-07 (Actual); Primary Completion 2020-08-04 (Actual); Study Completion 2020-08-04 (Actual)

PRIMARY OUTCOMES:
Epidemiologic data (Age and sex). | 400 days.
  Epidemiologic data (age rounded up in years, sex-number of males, females, and transgender, if any).
The Gross Motor Function Classification System (GMFCS) levels | 400 days
  The gross motor function of children with cerebral palsy was categorized into 5 different levels using the Gross Motor Function Classification System tool. A higher score means a worse condition.
The Modified Ashworth Scale (MAS) scores | 400 days
  The Modified Ashworth Scale (MAS) scores from 0 to 4 were used. A higher score means a worse condition.
Measurement of both Total and Unexplained cry durations | 400 days
  Caregivers measured both Total and Unexplained cry durations with a digital watch or a mobile phone in hours: minutes: seconds over five ten-day periods. MM1 while on placebo days 6-15 [P6-P15], and four measurements MM2 to MM5 while on treatment days 61-70 [T61-70], 241-250 [T241-250], 311-320 [T311-320], and 351-360 [T351-360].
  Statistician calculated means of cry duration in hours per day.

SECONDARY OUTCOMES:
Any other changes in the clinical profile observed during the study period and reported by the caregivers. | 400 days
  Any other changes in the clinical profile (frequency changes) observed during the study period were reported by the caregivers. The number and percentages of children with the change were calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Nagabhushana Rao Potharaju, BScMDDCHDM, Principal Investigator — Sathbhavana Brain Clinic, Hyderabad, India

IPD SHARING:
Plan to Share IPD: Yes
They must acknowledge the sharing.
Supporting Information: Study Protocol, SAP
Time Frame: One year
Access Criteria: For meta-analysis or a similar study

REFERENCES:
- [Background] Hagglund G, Burman-Rimstedt A, Czuba T, Alriksson-Schmidt AI. Self-versus Proxy-Reported Pain in Children with Cerebral Palsy: A Population-Based Registry Study of 3783 Children. J Prim Care Community Health. 2020 Jan-Dec;11:2150132720911523. doi: 10.1177/2150132720911523. PMID 32172660
- [Background] Ostojic K, Paget SP, Morrow AM. Management of pain in children and adolescents with cerebral palsy: a systematic review. Dev Med Child Neurol. 2019 Mar;61(3):315-321. doi: 10.1111/dmcn.14088. Epub 2018 Oct 31. PMID 30378122
- [Background] Parkinson KN, Dickinson HO, Arnaud C, Lyons A, Colver A; SPARCLE group. Pain in young people aged 13 to 17 years with cerebral palsy: cross-sectional, multicentre European study. Arch Dis Child. 2013 Jun;98(6):434-40. doi: 10.1136/archdischild-2012-303482. Epub 2013 Apr 20. PMID 23606716
- [Background] Fairhurst C, Shortland A, Chandler S, Will E, Scrutton D, Simonoff E, Baird G. Factors associated with pain in adolescents with bilateral cerebral palsy. Dev Med Child Neurol. 2019 Aug;61(8):929-936. doi: 10.1111/dmcn.14113. Epub 2018 Dec 3. PMID 30508224
- [Background] Alriksson-Schmidt A, Hagglund G. Pain in children and adolescents with cerebral palsy: a population-based registry study. Acta Paediatr. 2016 Jun;105(6):665-70. doi: 10.1111/apa.13368. Epub 2016 Mar 30. PMID 26880375
- [Background] Hauer J, Houtrow AJ; SECTION ON HOSPICE AND PALLIATIVE MEDICINE, COUNCIL ON CHILDREN WITH DISABILITIES. Pain Assessment and Treatment in Children With Significant Impairment of the Central Nervous System. Pediatrics. 2017 Jun;139(6):e20171002. doi: 10.1542/peds.2017-1002. PMID 28562301
- [Background] Westbom L, Rimstedt A, Nordmark E. Assessments of pain in children and adolescents with cerebral palsy: a retrospective population-based registry study. Dev Med Child Neurol. 2017 Aug;59(8):858-863. doi: 10.1111/dmcn.13459. Epub 2017 May 16. PMID 28509356
- [Background] Penner M, Xie WY, Binepal N, Switzer L, Fehlings D. Characteristics of pain in children and youth with cerebral palsy. Pediatrics. 2013 Aug;132(2):e407-13. doi: 10.1542/peds.2013-0224. Epub 2013 Jul 15. PMID 23858420
- [Background] Baxter P. Comorbidities of cerebral palsy need more emphasis--especially pain. Dev Med Child Neurol. 2013 May;55(5):396. doi: 10.1111/dmcn.12137. No abstract available. PMID 23574476
- [Background] Barney CC, Krach LE, Rivard PF, Belew JL, Symons FJ. Motor function predicts parent-reported musculoskeletal pain in children with cerebral palsy. Pain Res Manag. 2013 Nov-Dec;18(6):323-7. doi: 10.1155/2013/813867. PMID 24308022
- [Background] Ramstad K, Jahnsen R, Skjeldal OH, Diseth TH. Characteristics of recurrent musculoskeletal pain in children with cerebral palsy aged 8 to 18 years. Dev Med Child Neurol. 2011 Nov;53(11):1013-8. doi: 10.1111/j.1469-8749.2011.04070.x. PMID 22014321
- [Background] Ostojic K, Paget S, Kyriagis M, Morrow A. Acute and Chronic Pain in Children and Adolescents With Cerebral Palsy: Prevalence, Interference, and Management. Arch Phys Med Rehabil. 2020 Feb;101(2):213-219. doi: 10.1016/j.apmr.2019.08.475. Epub 2019 Sep 12. PMID 31521713
- [Background] Tedroff K, Gyllensvard M, Lowing K. Prevalence, identification, and interference of pain in young children with cerebral palsy: a population-based study. Disabil Rehabil. 2021 May;43(9):1292-1298. doi: 10.1080/09638288.2019.1665719. Epub 2019 Sep 17. PMID 31526138
- [Background] Voscopoulos C, Lema M. When does acute pain become chronic? Br J Anaesth. 2010 Dec;105 Suppl 1:i69-85. doi: 10.1093/bja/aeq323. PMID 21148657
- [Background] Blackman JA, Svensson CI, Marchand S. Pathophysiology of chronic pain in cerebral palsy: implications for pharmacological treatment and research. Dev Med Child Neurol. 2018 Sep;60(9):861-865. doi: 10.1111/dmcn.13930. Epub 2018 Jun 7. PMID 29882358
- [Background] Suter MR, Wen YR, Decosterd I, Ji RR. Do glial cells control pain? Neuron Glia Biol. 2007 Aug;3(3):255-68. doi: 10.1017/S1740925X08000100. PMID 18504511
- [Background] St James-Roberts I, Garratt R, Powell C, Bamber D, Long J, Brown J, Morris S, Dyson S, Morris T, Bhupendra Jaicim N. A support package for parents of excessively crying infants: development and feasibility study. Health Technol Assess. 2019 Oct;23(56):1-144. doi: 10.3310/hta23560. PMID 31597591
- [Background] Sacha GL, Foreman MG, Kyllonen K, Rodriguez RJ. The Use of Gabapentin for Pain and Agitation in Neonates and Infants in a Neonatal ICU. J Pediatr Pharmacol Ther. 2017 May-Jun;22(3):207-211. doi: 10.5863/1551-6776-22.3.207. PMID 28638303
- [Background] Asaro J, Robinson CA, Levy PT. Visceral Hyperalgesia: When to Consider Gabapentin Use in Neonates-Case Study and Review. Child Neurol Open. 2017 Feb 10;4:2329048X17693123. doi: 10.1177/2329048X17693123. eCollection 2017 Jan-Dec. PMID 28503628
- [Background] Bax M, Tydeman C, Flodmark O. Clinical and MRI correlates of cerebral palsy: the European Cerebral Palsy Study. JAMA. 2006 Oct 4;296(13):1602-8. doi: 10.1001/jama.296.13.1602. PMID 17018805
- [Background] Levine JD, Gordon NC, Fields HL. The mechanism of placebo analgesia. Lancet. 1978 Sep 23;2(8091):654-7. doi: 10.1016/s0140-6736(78)92762-9. PMID 80579
- [Background] Speyer R, Cordier R, Kim JH, Cocks N, Michou E, Wilkes-Gillan S. Prevalence of drooling, swallowing, and feeding problems in cerebral palsy across the lifespan: a systematic review and meta-analyses. Dev Med Child Neurol. 2019 Nov;61(11):1249-1258. doi: 10.1111/dmcn.14316. Epub 2019 Jul 22. PMID 31328797
- [Background] Calis EA, Veugelers R, Sheppard JJ, Tibboel D, Evenhuis HM, Penning C. Dysphagia in children with severe generalized cerebral palsy and intellectual disability. Dev Med Child Neurol. 2008 Aug;50(8):625-30. doi: 10.1111/j.1469-8749.2008.03047.x. PMID 18754902
- [Background] Samal P, Goyal V, Makharia GK, Das CJ, Gorthi SP, Y VV, Singh MB, Srivastava MVP. Transfer Dysphagia Due to Focal Dystonia. J Mov Disord. 2018 Sep;11(3):129-132. doi: 10.14802/jmd.17081. Epub 2018 Sep 30. PMID 30304925
- [Background] Li S, Shi S, Chen F, Lin J. The effects of baclofen for the treatment of gastroesophageal reflux disease: a meta-analysis of randomized controlled trials. Gastroenterol Res Pract. 2014;2014:307805. doi: 10.1155/2014/307805. Epub 2014 Oct 20. PMID 25389436